CLINICAL TRIAL: NCT06049329
Title: Investigation of Safety, Tolerability and Pharmacokinetic Properties of Multiple Doses of Oral NNC0487-0111 in Japanese Participants With Obesity
Brief Title: A Research Study of How a New Medicine Called Amycretin, Given as Tablets, Works in Japanese Men With Obesity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9487-5022; U1111-1284-5901 (Other: World Health Organization (WHO))
Record Dates: First submitted 2023-09-11; First posted 2023-09-22 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NNC0487-0111 (Experimental): Once-daily oral administration - 1 of 3 different doses
  Interventions: Drug: NNC0487-0111
- Placebo (Placebo Comparator): Once-daily oral administration - 1 of 3 different doses
  Interventions: Drug: Placebo (NNC0487-0111)

INTERVENTIONS:
Drug: NNC0487-0111 — Participants will get one tablet to swallow at the same time of the day.
  Arms: NNC0487-0111
Drug: Placebo (NNC0487-0111) — Participants will get one tablet to swallow at the same time of the day.
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate if a new study drug, NNC0487-0111, is safe and how it works in the participant's body, when given as an oral tablet to Japanese participants.

ELIGIBILITY:
Key inclusion criteria

* Male with both parents of Japanese descent
* Body mass index (BMI) between 25.0 and 34.9 kg/m^2 (both inclusive). Body weight equal to or greater than 65.0 kg
* Considered eligible based on the medical history, physical examination, and the results of vital signs, electrocardiogram (ECG) and clinical laboratory tests performed during the screening visit, as judged by the investigator

Key exclusion criteria

* Any disorder that in the investigator's opinion might jeopardise participant's safety or compliance with the protocol
* Presence of clinically significant gastrointestinal disorders or symptoms of gastrointestinal disorders potentially affecting absorption of drugs or nutrients, or as judged by the investigator

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-09-14 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events (TEAE) | From pre-dose on Day 1 until completion of the end of study visit Day 31
  Number of events

SECONDARY OUTCOMES:
AUC,MD; the area under the NNC0487-0111 plasma concentration-time curve after last multile dose | From pre-dose on Day 10 until Day 11 (24 hours post-dose)
  h*nmol/L
Cmax,MD; the maximum plasma concentration of NNC0487-0111 after last multiple dose | From pre-dose on Day 10 until completion of the end of study visit Day 31
  nmol/L
tmax,MD; the time of maximum plasma concentration of NNC0487-0111 after last multiple dose | From pre-dose on Day 10 until completion of the end of study visit Day 31
  hour

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Hakata Clinic, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: Yes
"According to the Novo Nordisk disclosure commitment on novonordisk-trials.com"
URL: http://novonordisk-trials.com